CLINICAL TRIAL: NCT01052558
Title: A Prospective, Randomized, Controlled, Parallel Groupos, Multicenter Clinical Investigation of the Glaukos Trabecular Micro-bypass Stent Model GTS400 in Conjunction With Cataract Surgery
Brief Title: GTS400 Stent Implantation in Conjunction With Cataract Surgery in Subjects With Open-angle Glaucoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Glaukos Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GC-006
Record Dates: First submitted 2010-01-13; First posted 2010-01-20 (Estimated); Last update posted 2015-05-19 (Estimated); Status verified 2015-05

CONDITIONS: Glaucoma
Keywords: Open angle; Glaucoma; Cataract; Surgery; Intraocular Pressure
MeSH Terms: conditions — Glaucoma; Cataract | interventions — Cataract Extraction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cataract Surgery Only (Active Comparator)
  Interventions: Procedure: Cataract Surgery
- Treatment with Cataract Surgery & Stents (Experimental): Ab interno trabecular micro-bypass stent surgery
  Interventions: Device: iStent Inject (GTS400)

INTERVENTIONS:
Device: iStent Inject (GTS400) — Subjects will be randomized to one of two groups. In this case, subjects will undergo cataract surgery with subsequent implantation of GTS400 stents.
  Other Names: Cataract surgery, stent implantation
  Arms: Treatment with Cataract Surgery & Stents
Procedure: Cataract Surgery — Subjects will be randomized to one of two groups. In this case, subjects will undergo cataract surgery only.
  Arms: Cataract Surgery Only

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of the GTS400 trabecular micro-bypass stent in reducing intraocular pressure (IOP) in subjects with open-angle glaucoma or ocular hypertension and co-existing cataract.

DETAILED DESCRIPTION:
Glaucoma is a collection of disorders characterized by progressive loss of visual field due to optic nerve damage. It is a leading cause of blindness in the United States, affecting 1-2% of individuals aged 60 and over. Management of glaucoma requires chronic, life-long treatment with a spectrum of therapeutic options including medications, laser treatment and surgical implants. The common goal among the various therapies is to lower intraocular pressure to target levels in order to prevent loss of visual fields from excessive pressure on the optic nerve.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with open-angle glaucoma in the study eye
* Subject must be on 1 to 3 glaucoma medications
* Subject able and willing to attend follow up visits for two years postop
* Subject able and willing to sign informed consent

Exclusion Criteria:

* Pseudoexfoliative and pigmentary glaucoma
* Prior glaucoma surgery of any type

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Actual)
Dates: Start 2010-01; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects with 12 month diurnalIOP </= 21 mmHg without use of ocular hypotensive medications for >/= 4 weeks prior to 12 month visit. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Jeff Wells, PharmD, MBA, Study Director — Glaukos Corporation; Jay Katz, MD, Study Chair — Wills Eye Institute; Thomas Jefferson University
Locations (22):
- United States (22):
  - Boozman-Hof Regional Eye Clinic, Rogers, Arkansas
  - North Bay Eye Associates, Inc., Petaluma, California
  - Glaucoma Consultants of Colorado, Parker, Colorado
  - The Center for Excellence in Eye Care, Miami, Florida
  - International Eye Center, Tampa, Florida
  - Clayton Eye Center / Eye Care Centers Management, Inc., Morrow, Georgia
  - Chicago Eye Specialists, Chicago, Illinois
  - Whitson Vision, PC, Indianapolis, Indiana
  - D'Ambrosio Eye Care, Lancaster, Massachusetts
  - Kresge Eye Institute, Detroit, Michigan
  - Discover Vision Centers, Independence, Missouri
  - Silverstein Eye Centers, Kansas City, Missouri
  - St. John's Medical Research Institute, Springfield, Missouri
  - Las Vegas Physician Research Group, Henderson, Nevada
  - Shepherd Eye Center, Las Vegas, Nevada
  - Ophthalmic Consultants of Long Island, Rockville Centre, New York
  - Thomas Mundorf, MD, Charlotte, North Carolina
  - Laurel Eye Clinic, Brookville, Pennsylvania
  - Carolina Eyecare Physicians, Mt. Pleasant, South Carolina
  - Vance Thompson Vision / Sanford Clinic, Sioux Falls, South Dakota
  - Texan Eye, Austin, Texas
  - Lehmann Eye Center, Nacogdoches, Texas